CLINICAL TRIAL: NCT06951191
Title: Applying a New Method for Pain Control in Intrauterine Device Insertion
Brief Title: Intrauterine Device Insertion Pain Management
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Kirby Woodall, Obstetrician/Gynecologist (MD), University of Missouri-Columbia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2101465
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: IUD Insertion Pain; IUD Insertion
Keywords: IUD; IUD insertion; IUD insertion pain; benzocaine; paracervical lidocaine; paracervical block
MeSH Terms: interventions — salicylhydroxamic acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo/Placebo (Placebo Comparator): Participants in this arm will receive saline spray and a needle stick without injection to the cervix
  Interventions: Other: Sham injection; Drug: Saline 0.9%
- Placebo/Lidocaine (Experimental): Participants in this arm will receive saline spray and injected lidocaine to the cervix
  Interventions: Drug: Lidocaine 2%; Drug: Saline 0.9%
- Benzocaine/Placebo (Experimental): Participants in this arm will receive benzocaine spray and a needle stick without injection to the cervix
  Interventions: Drug: Benzocaine 20%; Other: Sham injection
- Benzocaine/Lidocaine (Experimental): Participants in this arm will receive benzocaine spray and lidocaine injection to the cervix
  Interventions: Drug: Benzocaine 20%; Drug: Lidocaine 2%

INTERVENTIONS:
Drug: Benzocaine 20% — Benzocaine 20% topical spray
  Arms: Benzocaine/Lidocaine; Benzocaine/Placebo
Drug: Lidocaine 2% — Lidocaine 2% injectable solution
  Arms: Benzocaine/Lidocaine; Placebo/Lidocaine
Other: Sham injection — Sham injection to mimic Lidocaine paracervical block. Will use an injection needle and sham inject (no actual injection of fluid)
  Arms: Benzocaine/Placebo; Placebo/Placebo
Drug: Saline 0.9% — Saline spray to mimic use of benzocaine spray
  Arms: Placebo/Lidocaine; Placebo/Placebo

SUMMARY:
The goal of this clinical trial is to learn if use of topical benzocaine prior to the injection of lidocaine is effective in decreasing pain experienced during IUD insertion in patients 18 or older. The main question it aims to answer is:

Does topical use of benzocaine prior to lidocaine injection during IUD insertion effectively decrease pain experienced?

Researchers will compare benzocaine/lidocaine to benzocaine/placebo, placebo/lidocaine, and placebo/placebo to see if use of benzocaine prior to lidocaine injection works more effectively to decrease pain experienced rather than lidocaine, benzocaine, or placebo use alone.

Participants will:

* Arrive to clinic for previously scheduled IUD insertion
* Be screened, approached by research staff, and consented to join the trial
* Complete a demographic questionnaire
* Be randomly and blindly assigned to one of four groups
* Placebo/Placebo
* Placebo/Lidocaine
* Benzocaine/Placebo
* Benzocaine/Lidocaine
* All groups will be given 600mg of ibuprofen prior to procedure
* Be asked to rate their pain on a visual scale of 1-10 during several distinct points of the procedure.
* Be sent an optional survey to their email after the procedure

DETAILED DESCRIPTION:
The goal of the researchers is to determine if use of a topical benzocaine spray prior to lidocaine injection will cause a significant reduction in pain experienced by patients undergoing an IUD insertion. Participants will be screened, approached, and fully consented by research staff in the clinic prior to their IUD insertion. Demographics will be gathered from all participants through a questionnaire. All participants will be given 600mg of ibuprofen prior to the procedure, but will be randomized into one of 4 groups as to what interventions/placebos they will receive during their insertion. Interventions studied are benzocaine spray and lidocaine injection. Placebos will be saline spray and paracervical needle stick without injection. Participants will be asked to rate their pain on a visual scale of 1-10 at the following timepoints during the procedure:

* At the time of tenaculum placement
* At the time of uterine sounding
* At the time of IUD insertion and deployment
* Immediately after removal of instrumentation
* 15 minutes after the procedure Participants who provided an email will be sent an additional questionnaire to be responded to within 24 hours of the procedure. At the conclusion of the trial statistical analysis will be done to determine significance of pain reduction varying between the 4 groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing IUD insertion

Exclusion Criteria:

* IUD insertion <6 weeks postpartum
* Age <18 years
* Allergy or history of adverse effect of lidocaine, benzocaine (and inactive ingredients: flavor, isobutane, propane, polyethylene glycol, sodium saccharin), or ibuprofen
* Not undergoing IUD insertion
* Undergoing IUD insertion under general anesthesia
* Usage of anti-inflammatory or as-needed anxiety medications (not daily use) in the 12 hours prior to IUD insertion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean Pain Score During IUD Insertion Events as Quantified by Visual Analogue Scale | During IUD insertion procedure
  The Visual Analogue Scale (VAS) is a 0-10 pain intensity scale commonly used to assess pain intensity. Scores of 0 represent having no pain at all while scores of 10 represent worst pain possible; Therefore higher scores represent worse outcomes for pain management. VAS will be used to determine participant's levels of experienced pain at the 5 distinct events (tenaculum placement, uterine sounding, IUD insertion/deployment, immediately after instrumentation removal, 15 minutes post-procedure).

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri OB/GYN Associates-Smiley Lane, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Arm, Age, Parity, and Pain-scoring at different intervals
Supporting Information: Study Protocol
Time Frame: IPD will be made available via link after conclusion of study (anticipated by 12/31/2026) and will remain available indefinitely on the MOspace institutional repository so long as that service remains active.
Access Criteria: IPD will be made available to all through the use of the MOspace institutional repository. Individual participant data will be available on a spreadsheet detailing study arm, age, parity, and pain-scoring at the different intervals. This will be accessible through a unique URL that will be provided at the conclusion of the study and upon upload to the MOspace repository.